CLINICAL TRIAL: NCT05814965
Title: Association of Apical Periodontitis With Systemic Level of Inflammatory Markers : A Longitudinal Intervention Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dr. Sanjay Tewari 2023
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2; Apical Periodontitis
Keywords: Apical Periodontitis; Diabetes mellitus; High sensitivity C-reactive protein; Tumor necrosis factor-alpha; Interleukin; Glycated hemoglobin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periapical Periodontitis; Diabetes Mellitus | interventions — Endodontics

STUDY DESIGN:
Intervention Model Description: 280 patients 140 in DM (70 each with AP and 70 without AP) and 140 Systemically healthy (70 each with AP and 70 without AP)will be enrolled and compared for systemic markers .Subjects with AP will be provided Endodontics treatment and levels of markers will be assessed one year after Endodontics treatment. markers.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diabetic patients with Apical periodontitis (Experimental): Diabetic patients with Apical periodontitis received Endodontics treatment in form of Root canal treatment and assessment of inflammatory and metabolic markers
  Interventions: Procedure: endodontic treatment in the form of root canal treatment
- Healthy patients with Apical periodontitis (Experimental): systemically healthy participants patients with Apical periodontitis received Endodontics treatment in the form of root canal treatment and assessment of inflammatory markers
  Interventions: Procedure: endodontic treatment
- Diabetic patients with out Apical periodontitis (Active Comparator): systemic inflammatory markers along with metabolic markers will be assessed
  Interventions: Diagnostic Test: inflammatory markers will be assessed along with metabolic markers assessment
- Healthy participants without Apical periodontitis (Active Comparator): systemic inflammatory markers will be assessed
  Interventions: Diagnostic Test: assessment of inflammatory marker

INTERVENTIONS:
Procedure: endodontic treatment in the form of root canal treatment — Patients will receive endodontic treatment, and inflammatory markers will be assessed
  Other Names: RCT
  Arms: Diabetic patients with Apical periodontitis
Procedure: endodontic treatment — Patients will receive endodontic treatment in the form of root canal treatment, and inflammatory markers will be assessed along with metabolic markers assessment
  Arms: Healthy patients with Apical periodontitis
Diagnostic Test: assessment of inflammatory marker — assessment of inflammatory markers
  Arms: Healthy participants without Apical periodontitis
Diagnostic Test: inflammatory markers will be assessed along with metabolic markers assessment — inflammatory markers will be assessed along with metabolic markers assessment
  Arms: Diabetic patients with out Apical periodontitis

SUMMARY:
While cross-sectional studies have reported a significant association between diabetes and Apical Periodontics, prospective studies are scarce. This will be the first prospective interventional study to explore the cause-and-effect relation between AP and diabetes by assessment of levels of inflammatory markers in a longitudinal setting. Periapical healing in diabetics and nondiabetics will be compared after root canal treatment to evaluate the role of various physical and metabolic attributes on endodontic outcomes.

DETAILED DESCRIPTION:
This prospective longitudinal interventional study will be conducted on patients with radiographic evidence of AP in at least one teeth. Total of 280 patients will be selected from the pool of the patients referred to the Outpatient Department of Conservative Dentistry and Endodontics, Post Graduate Institute of Dental Sciences, Rohtak. They will be equally divided into two broad groups either without any systemic disease (140 patients) or with type 2 DM.(140 Patients with DM). Each group further divided into 70 patients with AP and 70 control in a systemically healthy group (selected to match participants in age, sex and BMI). Similarly,70 patients with AP and 70 control for participants with type 2 DM will be selected to additionally match with glycaemic control, drugs, and dietary measures apart from other physical attributes.

Analysis of systemic inflammatory markers IL-1b, IL-6, TNF- α and hsCRP will be done at baseline in both healthy and diabetic participants. Root canal treatment will be done in all the participants with AP and assessment of periapical healing and change in inflammatory markers will be done at 3, 6, and 12-month follow-up.

Sample size: Sample size was estimated based on the difference in hsCRP level in patients with AP and healthy control. Effect size of 0.52 was calculated based on the mean difference and pooled SD of 0.91 and 1.75 respectively. Sample size of 58 per group was obtained at 80% power and 0.05 alpha level. Anticipating 20% dropout, total 70 patients per group (in 4 groups total 280 patients)will be recruited.

Root Canal treatment Access opening will be done after rubber dam isolation and administration of local anesthesia.

debridement of the pulp chamber will be done and all canal orifices will be identified.

Negotiation of canals will be done. Working length will be determined using root ZX apex locator and will be verified radiographically. Root canal treatment will be performed with protaper rotary instrument using standard protocol. Coronal 2/3rd pre-enlargement will be performed with S1 and S2 files and apical third will be prepared with S1 followed by S2 and suitable finishing files depending on the size of apical binding file. Irrigation will be carried out using 5 mL of a 5% NaOCl solution between files. After preparation, the root canals will be irrigated with 5 mL 17% EDTA for 3 minutes to remove smear layer, followed by 5 mL 5% NaOCl. The final irrigation will be done with 5 mL distilled water. Intracanal dressing of Calcium hydroxide will be applied for 7 days and obturation of canal will be performed after 7 days on 2nd visit. The root canals will be dried using paper points and filled with laterally condensed gutta-percha (Dentsply Maillefer) and AH plus resin-after manipulation following manufacturers' instructions. Gutta- percha will be cut with a heated instrument and vertically condensed right at the orifice opening of the canals. Final composite resin restoration will be performed following manufacturer instruction. All the posterior teeth will be metal/ceramic crown after the completion of root canal treatment.

Follow up Follow-up and clinical and radiographic examinations will be carried out after every three months for one year. Glycaemic control in diabetes patients will also be evaluated by HbA1c values at each follow-up interval.

ELIGIBILITY:
Inclusion Criteria:

* Patients 30-55 year age group with minimum 20 natural teeth, with pulp necrosis confirmed by cold test and electric pulp test and radiographic evidence of periapical radiolucency with PAI score of ≥3 (24) or more in at least one mature tooth.
* control in the systemically healthy group will be selected to match participants in terms of age, sex, and BMI.
* control for participants with type 2 DM will be selected to additionally match with glycaemic control, drugs and dietary measures apart from other physical attributes.

Exclusion Criteria:

* Patients with clinical diagnosis of moderate to severe periodontitis (≥6 sites with probing depth ≥5 mm at separate teeth, with attachment loss and radiographic alveolar bone loss), Patients with immunosuppression, pregnancy, conditions requiring prophylactic antibiotics prior to dental treatment, bleeding disorders, medical conditions that may affect study participation (e.g., unstable cardiovascular disease) and chronic inflammatory conditions like rheumatoid

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-04-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
PAI SCORE | 12 MONTHS
  PERIAPICAL INDEX RADIOGRAPHIC EVALUATION
Interlukin 1B | 12 MONTHS
  INFLAMMATORY MARKER BY ELISA KIT
IL 6 | 12 MONTHS
  ESTIMATION OF NFLAMMATORY MARKER BY ELISA KIT
TNF -ALPHA | 12 MONTHS
  ESTIMATION OF NFLAMMATORY MARKER BY ELISA KIT
hs-CRP | 12 MONTHS
  ESTIMATION OF NFLAMMATORY MARKER BY ELISA KIT

CONTACTS AND LOCATIONS:
Overall Officials: SANJAY TEWARI, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES,ROHTAK
Locations (1):
- PGIDS, Rohtak, Haryana, India